CLINICAL TRIAL: NCT01871220
Title: Peri-implant Mucosa Dynamics Around Divergent and Concave Atlantis™ Abutment Transition Profiles.
Brief Title: Periimplant Mucosa Dynamics Around Divergent and Concave Atlantis Abutment Transition Profiles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Barwacz (Other)
Responsible Party: Sponsor-Investigator, Christopher Barwacz, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201302798
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Results first posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Dental Implant, Single-Tooth; Esthetics, Dental
Keywords: Implant Abutments; Oral Mucosa Changes; Implant Esthetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Divergent Abutment (Active Comparator): Divergent Transition Profile
  Interventions: Device: Divergent Transition Profile
- Concave Abutment (Experimental): Concave Transition Profile
  Interventions: Device: Concave Transition Profile

INTERVENTIONS:
Device: Concave Transition Profile — An Atlantis abutment is delivered with a concave transition profile.
  Arms: Concave Abutment
Device: Divergent Transition Profile — An Atlantis abutment is delivered with a linear transition profile
  Arms: Divergent Abutment

SUMMARY:
The purpose of this study is to compare the effect of two different implant abutment designs on gum tissue volume changes over time after implant placement.

DETAILED DESCRIPTION:
This is a randomized, prospective, controlled clinical trial comparing the facial gingival profiles around Atlantis™ abutments that have either a linear "divergent" or "concave" transitional profile on the facial and proximal aspect of the abutments.

Sixty study subjects requiring replacement of a single-rooted tooth with an implant-supported restoration will be recruited.

The Osseospeed™ Plus implant will be placed for all 60 subjects, with the use of Uni healing abutments to minimize lateral tissue displacement during healing. After implant placement, but before final impressions are obtained (8 weeks post-placement), subjects will be randomized to either a "divergent" or a "concave" transmucosal abutment design. For fabrication of the experimental abutment, Atlantis™ engineers will initially design a control "divergent" prototype that will be modified with a concavity on the facial and proximal transition zones to obtain an abutment that will otherwise retain all the features of the control abutment. Engineers will measure the linear topographical changes (ΔL=Lc-Ld) of the transition zone, as well as the volumetric change (x) on the mid-facial aspect of the abutment induced by the formation of a submucosal concavity. The primary outcome of the study will be the apico-coronal change of the peri-implant mucosal zenith from prosthesis delivery to one year.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* Subjects requiring replacement of a single-rooted tooth in the maxillary arch from first premolar to first premolar with an implant-supported restoration
* Teeth adjacent (mesial and distal) to study site must consist of two stable, natural teeth without signs of periodontal bone loss (<2.0mm) and/or significant soft tissue loss
* An opposing dentition with teeth, implants, or fixed prosthesis
* Subjects must be willing to follow instructions related to the study procedures
* Subjects must have read, understood, and signed the informed consent document

Exclusion Criteria:

Exclusion Criteria:

* Insufficient interocclusal space for implant placement and/or restoration at study site
* More than 2.0mm vertical bone loss at study site as measured from the mid-buccal crest of the bone on the adjacent teeth
* Untreated rampant caries
* Tobacco use free for ≤ 6 months
* Liver or kidney disfunction/failure
* Active severe infectious diseases that may affect normal healing and/or bone metabolism (e.g. AIDS)
* Uncontrolled diabetes
* Current alcohol or drug abuse
* Need for systemic corticosteroids or any other medication that would influence post-operative healing and/or osseointegration
* History of relevant head/neck cancer and/or radiation of the head/neck
* Subjects who currently use bisphosphonates or have a history of bisphosphonate use
* Subjects with metabolic bone diseases such as osteoporosis or Paget's disease of bone
* Known pregnancy or nursing mothers
* Unable or unwilling to return for follow-up visits for a period of 1 year
* Unlikely to be able to comply with study procedures according to investigators judgement

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-12-30 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A Barwacz, DDS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa College of Dentistry, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Divergent Abutment | Concave Abutment
Started | 29 | 32
Completed | 25 | 29
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Population: The baseline analysis population differs from the final results (i.e., 12 months after baseline), because 7 subjects were lost to follow-up over the course of the study, specifically 4 from the Divergent Allocation and 3 from the Concave Allocation.
Groups:
- Concave: Participants were missing a single-rooted tooth on the upper jaw and were randomly-assigned to receive a concave-shaped implant abutment.
- Divergent: Participants were missing a single-rooted tooth on the upper jaw and were randomly assigned to receive a divergent-shaped implant abutment.
- Total: Total of all reporting groups
Arm/Group | Concave | Divergent | Total
Number analyzed (Participants) | 32 | 29 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 26 | 52
  >=65 years | 6 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 10 | 29
  Male | 13 | 19 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Peri-Implant Mucosal Zenith Distance (in Millimeters) at the Concave/Divergent Abutment Sites
Description: Determine if there is a difference in soft tissue peri-implant zenith changes (in millimeters) for the concave/divergent abutment sites, specifically between at delivery and 1, 3, 6, and 12 months after Atlantis Abutment and Restoration Delivery. This measurement is taken using a standardized stereotactic digital photography system that allows for increased measurement accuracy and precision, specifically with the Canfield Dental Camera, Canfield Imaging Systems.
Time Frame: Delivery, and 1, 3, 6, and 12 months after Atlantis Abutment and Restoration Delivery
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Divergent Abutment | Concave Abutment
Number analyzed (Participants) | 25 | 29
millimeters
  Delivery | 9.860 (1.148) | 9.770 (1.146)
  1 Month After Delivery | 9.684 (1.203) | 9.618 (1.160)
  3 Months after Delivery | 9.674 (1.231) | 9.610 (1.174)
  6 Months after Delivery | 9.652 (1.166) | 9.599 (1.160)
  12 Months after Delivery | 9.622 (1.258) | 9.596 (1.167)

2. Secondary Outcome: Submarginal Buccal-lingual Thickness (Millimeters) in the Peri-implant Transition Zone Relative to a Fixed Reference Point After Prosthesis Delivery
Description: Determine if there is a difference in submarginal buccal-lingual soft tissue thickness in the peri-implant transition zone relative to a fixed reference point, specifically at baseline and 1, 3, 6, and 12 months after Atlantis Abutment and Restoration Delivery. This measurement is taken using a standardized stereotactic digital photography system that allows for increased measurement accuracy and precision, specifically with the Canfield Dental Camera, Canfield Imaging Systems.
Time Frame: Baseline and 1, 3, 6, and 12 months after Atlantis Abutment and Restoration Delivery
Population: The reason why the overall number of participants analyzed differs from the data in the rows is due to some participants being lost to follow-up.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Divergent Abutment | Concave Abutment
Number analyzed (Participants) | 27 | 31
millimeters
  Baseline | 2.722 (1.1294) | 2.814 (1.1291)
  1 month after delivery | 2.667 (0.6202) | 2.597 (0.6248)
  3 months after delivery: number analyzed (Participants) | 25 | 31
  3 months after delivery | 2.840 (0.7176) | 2.468 (0.5764)
  6 months after delivery: number analyzed (Participants) | 25 | 30
  6 months after delivery | 2.920 (0.6403) | 2.517 (0.5796)
  12 months after delivery: number analyzed (Participants) | 25 | 29
  12 months after delivery | 2.740 (0.7654) | 2.500 (0.5000)

3. Secondary Outcome: Keratinized Mucosa Width (Millimeters) at the Midfacial Aspect of the Implant Site.
Description: Determine if there is a difference in Keratinized Mucosa Width (millimeters) in the apico-coronal direction at the midfacial aspect of the implant site, specifically at baseline and 1, 3, 6, and 12 months after Atlantis Abutment and Restoration Delivery. This measurement is taken using a standardized stereotactic digital photography system that allows for increased measurement accuracy and precision, specifically with the Canfield Dental Camera, Canfield Imaging Systems.
Time Frame: Baseline and 1, 3, 6, and 12 months after Atlantis Abutment and Restoration Delivery
Population: The reason why the number analyzed in one or more rows differs from the overall number analyzed is that some subjects were lost to follow-up.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Divergent Abutment | Concave Abutment
Number analyzed (Participants) | 27 | 31
millimeters
  Baseline | 2.704 (1.1373) | 3.307 (1.8425)
  1 month after delivery | 3.407 (1.1522) | 3.936 (1.7212)
  3 months after delivery: number analyzed (Participants) | 25 | 31
  3 months after delivery | 3.620 (0.8930) | 4.177 (1.6711)
  6 months after delivery: number analyzed (Participants) | 25 | 30
  6 months after delivery | 3.478 (0.9946) | 4.067 (1.6439)
  12 months after delivery: number analyzed (Participants) | 25 | 29
  12 months after delivery | 3.560 (1.0832) | 4.035 (1.8609)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Divergent Abutment | Concave Abutment
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/32
Other Adverse Events (participants affected / at risk) | 0/29 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT01871220/Prot_SAP_000.pdf